CLINICAL TRIAL: NCT00814970
Title: The Complete® SE SFA Study: The Medtronic Complete Self-Expanding SFA Stent System for the Treatment of Atherosclerotic Lesions in the Superficial Femoral and/or Proximal Popliteal Arteries
Brief Title: The Complete® SE SFA Study for the Treatment of SFA/PPA Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Endovascular (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IP105; IDE G080143 (Other: FDA)
Record Dates: First submitted 2008-12-23; First posted 2008-12-25 (Estimated); Results first posted 2014-05-21 (Estimated); Last update posted 2016-04-13 (Estimated); Status verified 2016-02

CONDITIONS: Peripheral Vascular Disease
Keywords: PAD; peripheral arterial disease; stent; SFA; PPA
MeSH Terms: conditions — Peripheral Vascular Diseases; Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Complete SE Vascular Stent System (Experimental): COMPLETE SE Vascular Stent System - implantation of study device in native SFA and/or PPA for subjects with symptomatic ischemic peripheral arterial disease in the superficial femoral artery or proximal popliteal arteries with an occlusion or lesion greater or equal to 50 percent with lesions located above the knee and amenable to percutaneous treatment with angioplasty and vascular stent implantation.
  Interventions: Device: Complete SE Vascular Stent System

INTERVENTIONS:
Device: Complete SE Vascular Stent System — Complete SE Vascular Stent System in the treatment of de novo and/or restenotic lesions or occlusions in the Superficial Femoral Artery (SFA) and/or the Proximal Popliteal Artery (PPA) in subjects with symptomatic Peripheral Artery Disease (PAD).

SUMMARY:
To evaluate the safety and efficacy of the Complete SE SFA Stent System in the treatment of de novo and/or restenotic lesions or occlusions in the Superficial Femoral Artery (SFA) and/or Proximal Popliteal Artery (PPA) in subjects with symptomatic Peripheral Artery Disease (PAD).

DETAILED DESCRIPTION:
The Complete Self-Expanding (SE) SFA Stent is designed to be a permanent implant. It is cut from a nickel titanium alloy (Nitinol) tube and consists of a series of segments each connected to the next in a unique pattern to allow for flexibility and vessel conformability. Each segment consists of two struts and a crown (Figure 1). It is designed to produce optimal luminal diameter and increased scaffolding, and to maintain luminal patency.

ELIGIBILITY:
Inclusion Criteria:

1. Rutherford 2-4, with an occlusion or de novo and/or restenotic SFA/PPA lesion ≥50% and ankle-brachial index/toe-brachial index (ABI/TBI) <0.90/0.80.
2. Target lesion located at least 1 cm distal to the take-off of the profunda femoris artery and at least 3 cm proximal to the highest point of the cortical margin of the femur;
3. Target vessel reference diameter is ≥4.0 mm and ≤7.0 mm (visual estimate);
4. Target lesion length is ≥4.0 cm and ≤14.0 cm (visual estimate);
5. Adequate distal run-off to the ankle in the target limb (defined as having at least one patent calf vessel <50% stenosed;
6. Life expectancy >12 months.

   Exclusion Criteria:
7. Women who do not have a negative serum or urine pregnancy test documented within 7 days prior to enrollment;
8. Any condition that precludes safe access with percutaneous transluminal angioplasty (PTA) devices, such as: excessive peripheral artery disease, unresolved fresh thrombus in the target lesion/vessel, or a target lesion/vessel that is excessively tortuous or calcified;
9. Lesions in contralateral SFA/PPA that require intervention during the index procedure, or within 30 days before or after the index procedure;
10. Previous treatment to the target lesion within the 3 months prior to enrollment; previous femoropopliteal bypass in target vessel; previous stenting of the target lesion;
11. Target lesion located within an aneurysm or associated with an aneurysm in the vessel segment either proximal or distal to the target lesion;
12. Target lesion requires treatment other than standard PTA prior to stent placement (i.e., no other devices or procedures such as cutting balloons and laser atherectomy are permitted to be used during the index procedure);
13. History of bleeding diatheses or coagulopathy or will refuse blood transfusions;
14. Known impaired renal function, defined as creatinine >2.5 mg/dl;
15. Known platelet count <80,000 cells/mm3 or >700,000 cells/mm3;
16. Known white blood cell (WBC) of <3,000 cells/mm3;
17. Participation in another investigational device or drug study and has not completed the primary endpoint(s) or which clinically interferes with the Complete SE SFA Study endpoints, or previously enrolled in the Complete SE SFA Study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2008-11; Primary Completion 2011-09 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Laird, MD, Principal Investigator — University of California, Davis; Dierk Scheinert, PD, Principal Investigator — Park-Krankenhaus Leipzig-Sudost GmbH
Locations (4):
- United States (4):
  - Washington Hospital, Fremont, California
  - N. Florida Regional Medical Center, Gainesville, Florida
  - Munroe Regional Medical Center, Ocala, Florida
  - AnMed Health, Anderson, South Carolina

REFERENCES:
- [Derived] Laird JR, Jain A, Zeller T, Feldman R, Scheinert D, Popma JJ, Armstrong EJ, Jaff MR; Complete SE Investigators. Nitinol stent implantation in the superficial femoral artery and proximal popliteal artery: twelve-month results from the complete SE multicenter trial. J Endovasc Ther. 2014 Apr;21(2):202-12. doi: 10.1583/13-4548R.1. PMID 24754279

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was for a period of 20 months. Subjects were recruited at medical clinics who participate in clinical trials.
Groups:
- Complete Self-expanding (SE) Vascular Stent System: Device: Complete Self-expanding (SE) Vascular Stent System >
  > Complete Self-expanding (SE) Vascular Stent System: The Complete SE Vascular Stent System consists of a self-expanding stent and an over the wire (OTW) delivery system.
Period: Overall Study
Arm/Group | Complete Self-expanding (SE) Vascular Stent System
Started | 196
Completed | 146
Not Completed | 50

BASELINE CHARACTERISTICS:
Groups:
- Complete SE Vascular Stent System: Device: Complete SE Vascular Stent System>
  > Complete SE Vascular Stent System: The Complete SE Vascular Stent System consists of a self-expanding stent and an over the wire (OTW) delivery system.
Arm/Group | Complete SE Vascular Stent System
Number analyzed (Participants) | 196
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 74
  >=65 years | 122
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.7 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72
  Male | 124
Region of Enrollment [Number; unit: participants]
  United States | 133
  Germany | 48
  Belgium | 15

OUTCOME MEASURES:

1. Primary Outcome: Major Adverse Event (MAE) Rate
Description: Major Adverse Events (MAE) defined as device and/or procedure related death (or any death occurring post-procedure through Day 30), target limb loss and target lesion or target vessel revascularization.
Time Frame: 12 Months
Population: Intent-to-Treat Population
Measure: Number; unit: percentage of participants
Groups:
- Complete SE Vascular Stent System: Device: Complete SE Vascular Stent System >
  > Complete SE Vascular Stent System: The Complete SE Vascular Stent System consists of a self-expanding stent and an over the wire (OTW) delivery system.
Arm/Group | Complete SE Vascular Stent System
Number analyzed (Participants) | 196
percentage of participants | 11.0

2. Primary Outcome: Primary Patency Rate
Description: Primary patency defined as uninterrupted patency with no procedures performed on or at the margins of the treated segment, with no restenosis ≥ 50% as documented by peak systolic velocity ratio ≥2.0 as assessed by duplex ultrasound (DUS).
Time Frame: 12 Months
Population: Intention-to-Treat (ITT)
Measure: Number; unit: percentage of participants
Arm/Group | Complete SE Vascular Stent System
Number analyzed (Participants) | 196
percentage of participants | 72.6

3. Secondary Outcome: Major Adverse Event (MAE) Rate
Description: Major Adverse Events (MAE) defined as device and/or procedure related death (or any death occurring post-procedure through Day 30), target limb loss and target lesion or target vessel revascularization at the 30 day timepoint.
Time Frame: 30 days
Population: Intention-to-Treat (ITT)
Measure: Number; unit: percentage of participants
Arm/Group | Complete SE Vascular Stent System
Number analyzed (Participants) | 196
percentage of participants | 0.5

4. Secondary Outcome: Major Adverse Event (MAE) Rate
Description: Major Adverse Events (MAE) defined as device and/or procedure related death (or any death occurring post-procedure through Day 30), target limb loss and target lesion or target vessel revascularization at the 6 month timepoint.
Time Frame: 6 Months
Population: Intention-to-Treat (ITT)
Measure: Number; unit: percentage of participants
Arm/Group | Complete SE Vascular Stent System
Number analyzed (Participants) | 196
percentage of participants | 4.1

5. Secondary Outcome: Device Success
Description: The outcome is based on the angiographic evidence of <30% final residual stenosis of the target lesion using only the assigned device.
Time Frame: At time of deployment to the end of the treatment procedure (removal of vascular sheath from the patient).
Population: Intention-to-Treat (ITT)
Measure: Number; unit: percentage of lesions treated
Arm/Group | Complete SE Vascular Stent System
Number analyzed (Participants) | 196
percentage of lesions treated | 90.0

6. Secondary Outcome: Lesion Success
Description: The outcome is based on the angiographic evidence of <30% final residual stenosis of the target lesion using either the Complete SE SFA Stent System or other standard percutaneous devices.
Time Frame: At time of deployment to the end of the treatment procedure (removal of vascular sheath from the patient).
Population: Intention-to-Treat (ITT)
Measure: Number; unit: percentage of lesions treated
Arm/Group | Complete SE Vascular Stent System
Number analyzed (Participants) | 196
percentage of lesions treated | 90.0

7. Secondary Outcome: Procedure Success
Description: The outcome is based on the angiographic evidence of <30% final residual stenosis of the target lesion after stent implantation and no occurrence of a procedure-related Major Adverse Events (MAE) prior to hospital discharge.
Time Frame: At time of deployment to time of hospital discharge
Population: Intention-to-Treat (ITT)
Measure: Number; unit: percentage of lesions treated
Arm/Group | Complete SE Vascular Stent System
Number analyzed (Participants) | 196
percentage of lesions treated | 89.1

8. Secondary Outcome: Assisted Primary Patency
Description: Defined as vessel patency resulting from a procedure performed in the treated segment.
Time Frame: 12 months
Population: Intention-to-Treat (ITT)
Measure: Number; unit: percentage of participants
Arm/Group | Complete SE Vascular Stent System
Number analyzed (Participants) | 196
percentage of participants | 78.3

9. Secondary Outcome: Secondary Patency Rate
Description: Defined as vessel patency resulting from any procedure that restores patency.
Time Frame: 12 Months
Population: Intention-to-Treat (ITT)
Measure: Number; unit: percentage of participants
Arm/Group | Complete SE Vascular Stent System
Number analyzed (Participants) | 196
percentage of participants | 78.9

10. Secondary Outcome: Change in Quality of Life - Improvement in Rutherford Class by >= 1 Category
Description: Improvement in Rutherford class by ≥ 1 category increase at 12 months from pre-procedure according to the Rutherford Scale Classification. The Rutherford Classification is a categorical scale (0 - 6) used by clinicians to assess the degree of peripheral arterial disease in a person. The scale begins with 0 (no symptoms) and ends with 6 (worse case symptoms).
Time Frame: 12 months
Population: Intention-to-Treat (ITT)
Measure: Number; unit: percentage of participants
Arm/Group | Complete SE Vascular Stent System
Number analyzed (Participants) | 196
percentage of participants | 90.9

11. Secondary Outcome: Change in Quality of Life - Increase in Ankle-brachial Index (ABI) or Toe-brachial Index (TBI) >= 0.15
Description: Increase in ABI/TBI ≥ 0.15 at 12 months from pre-procedure. An increase in ABI/TBI of 0.15 or greater is considered by clinicians to be a significant improvement.
Time Frame: 12 Months
Population: Intention-to-Treat (ITT)
Measure: Number; unit: percentage of participants
Arm/Group | Complete SE Vascular Stent System
Number analyzed (Participants) | 196
percentage of participants | 64.5

12. Secondary Outcome: Change in Quality of Life - Decrease in Rutherford Class >= 1 Category
Description: Decline in Rutherford class ≥ 1 category at 30 days when compared to pre-procedure according to the Rutherford Scale Classification. The Rutherford Classification is a categorical scale (0 - 6) used by clinicians to assess the degree of peripheral arterial disease in a person. The scale begins with 0 (no symptoms) and ends with 6 (worse case symptoms).
Time Frame: 30 Days
Population: Intention-to-Treat (ITT)
Measure: Number; unit: percentage of participants
Arm/Group | Complete SE Vascular Stent System
Number analyzed (Participants) | 196
percentage of participants | 89.7

13. Secondary Outcome: Percentage of Participants Free From Strut Fractures
Description: Defined as percent free from strut fractures. Percentage based on number of stents implanted with flat plate x-ray follow-up.
Time Frame: 12 Months
Population: Intention-to-Treat (ITT)
Measure: Number; unit: percentage of participants
Units Other Than Participants: Stents implanted with x-ray follow-up
Arm/Group | Complete SE Vascular Stent System
Number analyzed (Participants) | 196
Number analyzed (Stents implanted with x-ray follow-up) | 189
percentage of participants | 100.0

14. Secondary Outcome: Clinically-driven Target Lesion Revascularization (TLR) Rate
Description: Defined as those revascularizations in which the subject has ischemic symptoms consistent with changes within the target lesion as demonstrated by: a change (decrease from post-procedure) in the Rutherford scale by at least one category, or a change (decrease from post-procedure) in ABI/TBI >= 0.15
Time Frame: 12 Months
Population: Intention-to-Treat (ITT)
Measure: Number; unit: percentage of participants
Arm/Group | Complete SE Vascular Stent System
Number analyzed (Participants) | 196
percentage of participants | 8.4

15. Secondary Outcome: Major Adverse Event (MAE) Rate
Description: Major Adverse Events (MAE) defined as device and/or procedure related death (or any death occurring post-procedure through Day 30), target limb loss and target lesion or target vessel revascularization at the 24 month timepoint.
Time Frame: 24 Months
Population: Intention-to-Treat
Measure: Number; unit: percentage of participants
Arm/Group | Complete SE Vascular Stent System
Number analyzed (Participants) | 196
percentage of participants | 22.5

16. Secondary Outcome: Percentage of Participants Free From Strut Fractures
Description: Defined as percent free from strut fractures. Percentage based on number of stents implanted with flat plate x-ray follow-up at the 24 month timepoint.
Time Frame: 24 Months
Population: Intention-to-Treat (ITT)
Measure: Number; unit: percentage of participants
Units Other Than Participants: Stents implanted with x-ray follow-up
Arm/Group | Complete Self-expanding (SE) Vascular Stent System
Number analyzed (Participants) | 196
Number analyzed (Stents implanted with x-ray follow-up) | 159
percentage of participants | 100.0

17. Secondary Outcome: Major Adverse Event (MAE) Rate
Description: Major Adverse Events (MAE) defined as device and/or procedure related death (or any death occurring post-procedure through Day 30), target limb loss and target lesion or target vessel revascularization at the 36 month timepoint.
Time Frame: 36 Months
Population: Intention-to-Treat
Measure: Number; unit: percentage of participants
Arm/Group | Complete SE Vascular Stent System
Number analyzed (Participants) | 196
percentage of participants | 30.2

18. Secondary Outcome: Percentage of Participants Free From Strut Fractures
Description: Defined as percent free from strut fractures. Percentage based on number of stents implanted with flat plate x-ray follow-up at the 36 month timepoint.
Time Frame: 36 Months
Population: Intention-to-Treat
Measure: Number; unit: percentage of participants
Units Other Than Participants: Stents implanted with x-ray follow-up
Arm/Group | Complete SE Vascular Stent System
Number analyzed (Participants) | 196
Number analyzed (Stents implanted with x-ray follow-up) | 159
percentage of participants | 100.0

ADVERSE EVENTS:
Time Frame: 12 months
Groups:
- 1. Complete SE Vascular Stent System: Complete SE Vascular Stent System: The Complete SE Vascular Stent System consists of a self-expanding stent and an over the wire (OTW) delivery system.
Arm/Group | 1. Complete SE Vascular Stent System
Serious Adverse Events (participants affected / at risk) | 117/196
Other Adverse Events (participants affected / at risk) | 50/196
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1. Complete SE Vascular Stent System (N=196)
Anaemia (Blood and lymphatic system disorders) | 8 (9)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Acute Myocardial Infarction (Cardiac disorders) | 4 (4)
Angina Pectoris (Cardiac disorders) | 4 (4)
Angina Unstable (Cardiac disorders) | 3 (3)
Atrial Fibrillation (Cardiac disorders) | 4 (4)
Atrioventricular Block (Cardiac disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Cardiac Failure (Cardiac disorders) | 3 (4)
Cardiac Failure Congestive (Cardiac disorders) | 3 (4)
Coronary Artery Disease (Cardiac disorders) | 10 (10)
Myocardial Infarction (Cardiac disorders) | 2 (2)
Myocardial Ischaemia (Cardiac disorders) | 1 (1)
Sick Sinus Syndrome (Cardiac disorders) | 2 (2)
Ventricular Tachycardia (Cardiac disorders) | 2 (2)
Gastrointestinal Angiodysplasia (Congenital, familial and genetic disorders) | 1 (1)
Vitreous Haemorrhage (Eye disorders) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Abdominal Strangulated Hernia (Gastrointestinal disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Duodenal Ulcer Perforation (Gastrointestinal disorders) | 1 (1)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 3 (3)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1 (1)
Mesenteric Vein Thrombosis (Gastrointestinal disorders) | 1 (1)
Pancreatitis Acute (Gastrointestinal disorders) | 2 (2)
Small Intestinal Obstruction (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1)
Asthenia (General disorders) | 1 (2)
Catheter Site Haemorrhage (General disorders) | 1 (1)
Chest Pain (General disorders) | 9 (9)
Gait Disturbance (General disorders) | 2 (2)
Impaired Healing (General disorders) | 2 (2)
Non-Cardiac Chest Pain (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Vessel Puncture Site Haematoma (General disorders) | 1 (1)
Wound Necrosis (General disorders) | 1 (1)
Bile Duct Stone (Hepatobiliary disorders) | 1 (2)
Gallbladder Disorder (Hepatobiliary disorders) | 1 (1)
Bronchitis (Infections and infestations) | 4 (4)
Bronchopneumonia (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 4 (5)
Clostridium Difficile Colitis (Infections and infestations) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1)
Gangrene (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Lobar Pneumonia (Infections and infestations) | 1 (1)
Localised Infection (Infections and infestations) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1)
Osteomyelitis Acute (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 5 (5)
Sepsis (Infections and infestations) | 5 (5)
Subcutaneous Abscess (Infections and infestations) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 2 (4)
Wound Infection (Infections and infestations) | 1 (1)
Device Electrical Finding (Injury, poisoning and procedural complications) | 1 (1)
Hip Fracture (Injury, poisoning and procedural complications) | 1 (1)
Humerus Fracture (Injury, poisoning and procedural complications) | 1 (1)
In-Stent Arterial Restenosis (Injury, poisoning and procedural complications) | 14 (15)
Pelvic Fracture (Injury, poisoning and procedural complications) | 1 (1)
Stent Occlusion (Injury, poisoning and procedural complications) | 5 (5)
Diabetes Mellitus (Metabolism and nutrition disorders) | 1 (1)
Failure To Thrive (Metabolism and nutrition disorders) | 1 (1)
Gout (Metabolism and nutrition disorders) | 1 (1)
Metabolic Acidosis (Metabolism and nutrition disorders) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 2 (3)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Carotid Artery Stenosis (Nervous system disorders) | 7 (8)
Cerebral Infarction (Nervous system disorders) | 1 (1)
Cerebrovascular Accident (Nervous system disorders) | 2 (2)
Dizziness (Nervous system disorders) | 1 (2)
Hemiparesis (Nervous system disorders) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1)
Spinal Claudication (Nervous system disorders) | 1 (1)
Transient Ischaemic Attack (Nervous system disorders) | 1 (1)
Alcohol Withdrawal Syndrome (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Mental Status Changes (Psychiatric disorders) | 2 (2)
Psychotic Disorder (Psychiatric disorders) | 1 (1)
Renal Artery Stenosis (Renal and urinary disorders) | 1 (1)
Renal Failure Acute (Renal and urinary disorders) | 4 (4)
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Skin Ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Hip Arthroplasty (Surgical and medical procedures) | 1 (1)
Peripheral Revascularisation (Surgical and medical procedures) | 3 (3)
Tendon Sheath Incision (Surgical and medical procedures) | 1 (1)
Wound Debridement (Surgical and medical procedures) | 1 (1)
Aneurysm (Vascular disorders) | 1 (1)
Arterial Occlusive Disease (Vascular disorders) | 2 (2)
Arterial Restenosis (Vascular disorders) | 2 (2)
Arterial Stenosis (Vascular disorders) | 1 (3)
Arterial Stenosis Limb (Vascular disorders) | 5 (5)
Artery Dissection (Vascular disorders) | 7 (7)
Femoral Arterial Stenosis (Vascular disorders) | 16 (17)
Femoral Artery Occlusion (Vascular disorders) | 3 (3)
Haematoma (Vascular disorders) | 1 (1)
Iliac Artery Stenosis (Vascular disorders) | 1 (1)
Intermittent Claudication (Vascular disorders) | 13 (15)
Peripheral Arterial Occlusive Disease (Vascular disorders) | 2 (2)
Peripheral Artery Dissection (Vascular disorders) | 3 (3)
Peripheral Embolism (Vascular disorders) | 1 (1)
Peripheral Ischaemia (Vascular disorders) | 3 (3)
Peripheral Vascular Disorder (Vascular disorders) | 1 (1)
Vascular Pseudoaneurysm (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1. Complete SE Vascular Stent System (N=196)
Chest Pain (General disorders) | 12 (13)
Back Pain (Musculoskeletal and connective tissue disorders) | 16 (16)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 15 (18)
Intermittent Claudication (Vascular disorders) | 17 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days